CLINICAL TRIAL: NCT03655457
Title: Evaluation of the Efficacy of Different Surfactant Preparations in Preterm Infants by Lung Ultrasound
Brief Title: Evaluation of the Efficacy of Surfaktant in Preterm Infants by Lung Ultrasound
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zekai Tahir Burak Women's Health Research and Education Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 22032018
Record Dates: First submitted 2018-03-22; First posted 2018-08-31 (Actual); Last update posted 2018-12-11 (Actual); Status verified 2018-03

CONDITIONS: Lung Ultrasound Scores
Keywords: Lung; RDS; Surfaktant

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group 1 Poractant alfa (Experimental): Poractant alfa generic name: curosurf 120 and 240 mg flk dosage: 200 mg/ kg intratracheal application frequency and duration: in the first two hours
  Interventions: Device: group 1 Poractant alfa
- group 2 beractant (Active Comparator): beractant generic name: survanta 8 cc flk dosage: 4 cc/ kg intratracheal application frequency and duration: in the first two hours
  Interventions: Device: group 2 beractant

INTERVENTIONS:
Device: group 1 Poractant alfa — Comparison of lung usg scores in infants treated with Poractant alfa and Beractant: 0 indicates A-pattern (defined by the presence of the only A-lines); 1, B-pattern (defined as the presence of ≥3 well-spaced B-lines); 2, severe B-pattern (defined as the presence of crowded and coalescent B-lines with or without consolidations limited to the subpleural space); and 3, extended consolidations.
  Arms: group 1 Poractant alfa
Device: group 2 beractant — lComparison of lung usg scores in infants treated with Poractant alfa and Beractant: 0 indicates A-pattern (defined by the presence of the only A-lines); 1, B-pattern (defined as the presence of ≥3 well-spaced B-lines); 2, severe B-pattern (defined as the presence of crowded and coalescent B-lines with or without consolidations limited to the subpleural space); and 3, extended consolidations.
  Arms: group 2 beractant

SUMMARY:
To compare the lung ultrasound scores after two different natural surfactant administration as a parameter reflecting lung inflation. Poractant alfa decreases lung ultrasound scores as efficient as beractant treatment

DETAILED DESCRIPTION:
Outcomes:

Improvement of Lung usg scores after surfactanct and the difference between groups at different time points (2nd and 6hr).

Secondary outcome:

The correlation between lung usg scores and clinical scores (silverman scores), FiO2 and PCO2 levels, failure of weaning to noninvasive ventilation after surfactant Preterm infants of 32 gestational weeks and below, who admit to the NICU with signs of respiratory distress, treated with non invasive or mechanical ventilation and require surfactant treatment in 6 hours of life will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Preterm infants of 32 gestational weeks and below, who admit to the NICU with signs of respiratory distress, treated with non invasive or mechanical ventilation and require surfactant treatment in 6 hours of life will be enrolled.

Exclusion Criteria:

* major congenital anomalies.

Ages: 1 Hour to 6 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 64 (Estimated)
Dates: Start 2018-03-21 (Actual); Primary Completion 2019-01-30 (Estimated); Study Completion 2019-02-28 (Estimated)

PRIMARY OUTCOMES:
Lung usg scores | first days
  Evaluation of Lung Usg Scores in infants treated with surfactant in the first six hours (Brat lung usg scores). Each item scored 0-3. (0 indicates A-pattern (defined by the presence of the only A-lines); 1, B-pattern (defined as the presence of ≥3 well-spaced B-lines); 2, severe B-pattern (defined as the presence of crowded and coalescent B-lines with or without consolidations limited to the subpleural space); and 3, extended consolidations.)
  - Higher values represent a worse outcome

CONTACTS AND LOCATIONS:
Overall Officials: Evrim Alyamaç Dizdar, MD, Study Director — zekai tahir burak matarnity teaching hospital
Locations (1):
- Zekai Tahir Burak Matarnity Teaching, Ankara, Turkey (Türkiye)